CLINICAL TRIAL: NCT02882789
Title: A Randomized, Single Blind, Single Dose, Phase I Study to Investigate the Pharmacokinetics, Safety, and Tolerability of Intravenous Dosage Form of LCB01-0371 in Healthy Male Volunteers
Brief Title: IV Dosage Form of LCB01-0371 Phase I Study in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: LigaChem Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LCB01-0371-16-1-01
Record Dates: First submitted 2016-08-09; First posted 2016-08-30 (Estimated); Last update posted 2018-04-10 (Actual); Status verified 2017-03

CONDITIONS: Healthy
MeSH Terms: interventions — delpazolid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- LCB01-0371 200mg (Experimental): LCB01-0371 IV 200 mg
  Interventions: Drug: LCB01-0371
- LCB01-0371 400mg (Experimental): LCB01-0371 IV 400 mg
  Interventions: Drug: LCB01-0371; Drug: LCB01-0371 400mg
- LCB01-0371 800mg (Experimental): LCB01-0371 IV 800 mg
  Interventions: Drug: LCB01-0371

INTERVENTIONS:
Drug: LCB01-0371 — Cohort1 & 3: Placebo-controlled, Single ascending dose administration
  Other Names: LCB01-0371 or placebo
Drug: LCB01-0371 400mg — Cohort 2: Crossover designed administration
  Other Names: LCB01-0371 400mg 2 tablet
  Arms: LCB01-0371 400mg

SUMMARY:
Primary - To investigate the Pharmacokinetics, Safety, and Tolerability of Intravenous dosage form of LCB01-0371 comparing to oral dosage in Healthy Male Volunteers Secondary

• To investigate the absolute bio availability of LCB01-0371 after a single intravenous dose

ELIGIBILITY:
Inclusion Criteria:

1. Healthy Male between 19 and 39 years of age at the time of screening
2. Subjects with body mass index (BMI) between 19 and 27 at the time of screening
3. Agree to continue to use a medically reliable dual contraception and not to donate sperm until 28 days of study completion
4. Capable of giving written informed consent, willing to participate in this clinical trial, and willing to comply with all study requirements

Exclusion Criteria:

1. History of gastrointestinal problem (e.g. Crohn's disease, gastro-intestinal ulcer) which is affect to absorption OR surgical history except appendectomy, herniotomy
2. History of allergy, cardiovascular, peripheral vascular, skin, mucous membrane, eyes, otorhinolaryngologic, respiratory, musculoskeletal, infectious disease, gastroenterologic, liver, billiary, endocrinologic, kidney, genitourinary, neuropsychiatric, hemato-oncologic problem(s) or fracture etc.

Ages: 19 Years to 39 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
To assess Peak Plasma Concentration(Cmax) of LCB01-0371 | through study completion per patient, an average of 8 days (+ - 1 D)

CONTACTS AND LOCATIONS:
Locations (1):
- Bae KS, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Cho YS, Lim HS, Han S, Yoon SK, Kim H, Cho YL, Nam HS, Bae KS. Single-dose Intravenous Safety, Tolerability, and Pharmacokinetics and Absolute Bioavailability of LCB01-0371. Clin Ther. 2019 Jan;41(1):92-106. doi: 10.1016/j.clinthera.2018.11.009. Epub 2018 Dec 15. PMID 30559004